CLINICAL TRIAL: NCT05595239
Title: The Efficacy of Different Mode of Blood Purification in Septic Children
Brief Title: Blood Purification in Septic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other); Shandong Provincial Hospital (Other Government); Children's Hospital of Soochow University (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: fdpicu-26
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Blood Purification
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard treatment+CVVH (Experimental)
  Interventions: Device: blood purification(CVVH)
- standard treatment+TPE+CVVH (Experimental)
  Interventions: Device: blood purification(TPE+CVVH)
- standard treatment+HP+CVVH (Experimental)
  Interventions: Device: blood purification(HP+CVVH)

INTERVENTIONS:
Device: blood purification(CVVH) — After the sepsis patients were enrolled, they were treated with blood purification in CVVH mode, 24 hours per day, for 3 consecutive days
  Arms: standard treatment+CVVH
Device: blood purification(TPE+CVVH) — After the sepsis patients were enrolled, they were treated with blood purification in TPE mode 2 hours at first and then in CVVH mode 22 hours in the first two days, and then in CVVH mode 24 hours
  Arms: standard treatment+TPE+CVVH
Device: blood purification(HP+CVVH) — After the sepsis patients were enrolled, they were treated with blood purification in HP mode 2 hours at first and then in CVVH mode 22 hours in the first two days, and then in CVVH mode 24 hours
  Arms: standard treatment+HP+CVVH

SUMMARY:
In septic shock, dysregulated host responses to pathogens lead to cytokine storms that damage host tissues and organs, further contributing to the development of organ dysfunction and increased mortality. For sepsis, blood purification can remove inflammatory factors in sepsis by filtration or adsorption, so as to achieve the purpose of reducing inflammatory mediators in the body. However, there are few prospective randomized controlled studies in children. Therefore, this study intends to compare the efficacy and prognosis of different blood purifications on children with sepsis through randomized controlled studies, so as to provide a corresponding basis for the treatment of children with sepsis blood purification.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction resulting from a dysregulated host response to infection. In septic shock, dysregulated host responses to pathogens lead to cytokine storms that damage host tissues and organs, further contributing to the development of organ dysfunction and increased mortality.

Blood purification therapy is gradually developed on the basis of renal replacement therapy, and now it is more and more widely used in the field of critical care in children. The main mechanisms are divided into dispersion, convection and adsorption. For sepsis, in addition to using the convection mechanism to remove the inflammatory mediators in the middle molecules, there are many adsorption membranes or adsorption columns used to adsorb the inflammatory factors in sepsis, so as to achieve the purpose of reducing the inflammatory mediators in the body. CVVH, HP and TPE can reduce the level of inflammation in the body in different ways, but the results of reducing inflammatory factors are different, and the outcomes of patients are also different.

Blood purification treatment can reduce inflammatory mediators in sepsis, but there are few prospective randomized controlled studies in children. Therefore, this study intends to compare the efficacy and prognosis of different blood purification in children with sepsis through a randomized controlled study. Provide the corresponding basis for blood purification treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Meet the 2005 diagnostic criteria for sepsis
* Age 29 days - 18 years old
* Sepsis-induced dysfunction of more than one organ or abnormal tissue perfusion, or septic shock
* Diagnosis < 48 hours

Exclusion Criteria:

* Inability to obtain an informed consent from the subject, family member or an authorized surrogate
* Subject has end-stage renal disease and requires chronic dialysis
* There is clinical support for non-septic shock
* Subject has had chest compressions as part of cardiopulmonary resuscitation this hospitalization without immediate return to communicative state
* Subject has uncontrolled hemorrhage
* Subject has immunodeficiency diseases
* Subject has received chemoradiotherapy or immunosuppressive therapy in the 14 days before enrollment
* HIV infection in association with a last known or suspected CD4 count of <50/mm3
* Subject has sustained extensive third-degree burns within the past 7 days
* Subject has known sensitivity or allergy to heparin or has a history of heparin associated thrombocytopenia
* Subject is currently enrolled in an investigational drug or device trial
* Subject has been previously enrolled in the current trial
* Any other condition, that in the opinion of the investigator, would preclude the subject from being a suitable candidate for enrollment, such as end stage chronic illness with no reasonable expectation of survival to hospital discharge
* Known hypersensitivity to hemofilter
* Subject has received organ transplantation
* Subject is expected to die within 24 hours

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cytokine change | from enrollment to the 3th days
  This is a binary variable. It is also a compositional variable including IL-6, IL-10, TNF-a, IL-4, IL-2 and etc. If one of the factors changes, it is considered that the variable changes. If the cytokine drops below half of the original value, it is considered to be changed. The cytokine would be measured measured at the 7th day after enrollment
organ injury changes | from enrollment to the 3th days
  the difference of the organ injury changes would be measured at the 3th day after enrollment

SECONDARY OUTCOMES:
survival rate | from enrollment to the 28th days
  the survival rate would be measured at the 28th day after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Lu Guoping, Shanghai, Shanghai Municipality, China